CLINICAL TRIAL: NCT00134615
Title: Testing the Right Question Project Health Education Strategy in a Mental Health Setting
Brief Title: Testing the Right Question Project (RQP) Health Education Strategy in a Mental Health Setting
Acronym: RQP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Margarita Alegria, PhD, Chief, Disparities Research Unit, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CHA-IRB-0080/07/04; P20MD000537 (NIH)
Record Dates: First submitted 2005-08-24; First posted 2005-08-25 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Diagnosis, Psychiatric
Keywords: decision-making; patient activation; empowerment; mental health; Depression; Anxiety; Other Psychiatric Disorder
MeSH Terms: conditions — Mental Disorders; Patient Participation; Empowerment; Psychological Well-Being; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- RQP-MH (Experimental): These participants receive the RQP-MH intervention
  Interventions: Behavioral: RQP patient health education module

INTERVENTIONS:
Behavioral: RQP patient health education module

SUMMARY:
The purpose of this pilot project is to test the effectiveness of three 20 minute health education modules on patient empowerment, patient activation and retention in care.

DETAILED DESCRIPTION:
Recent research has demonstrated positive outcomes for patients who take an active role in their mental health care (Linhorst & Eckert, 2003). Patients who participate in the decision-making process are more satisfied with services, have a greater sense of self-efficacy and confidence, an increased ability to cope with daily life, and are more likely to achieve their treatment goals (Linhorst & Eckert, 2003). As defined by Chamberlin and Schene (1997), empowerment in mental health care requires having access to information and resources, having a range of options from which to make choices, learning to think critically, and having the power to make decisions. Cooper-Patrick et al. (1999) indicate that minority patients are less likely to have a collaborative relationship with providers than are otherwise similar white patients. Thus, there is a need for minority patients to learn to take a more active role in their care. One way to address the need for increased empowerment and activation among minority mental health patients is to provide them with training to enhance their communication and decision-making skills. The Right Question Project (RQP) is a consumer educational technique designed for this purpose and developed for use in multiple settings. The proposed study will examine the effectiveness of RQP with a Latino population.

The Right Question Project (RQP) is a non-profit organization that works primarily with low- and moderate-income communities with a history of disengagement from education, health care, and other social services. The RQP approach differs from traditional models of client empowerment in that instead of supplying clients with solutions to problems, the RQP gives them a means to develop their own solutions. RQP teaches clients to identify important issues, formulate questions, and devise plans to communicate and act in effective ways that address factors impacting their health. The RQP methodology involves:

* establishing a set of beliefs, principles, and values about client involvement;
* teaching a skill-building technique that helps clients to think critically and ask the "right" questions, leading to the answers they need; and
* giving clients a framework to create action plans and use their question-formulation skills.

The RQP methodology is designed to build a permanent skill that clients can apply in health care, as well as in other contexts that involve self-advocacy (e.g., getting better child care). Thus far, implementation of the Right Question Project has shown that clients of any education or literacy level can easily participate and benefit from the methodology's three-step approach. RQP has been particularly successful in educational settings (Cohen, 1995).

The focus of the RQP health education module is to help patients learn how to formulate and ask questions of their health care providers, in order to improve the quality of their care. The Right Question Project, Inc. developed this protocol and trained staff at the Cambridge Health Alliance (CHA) to conduct health education modules with psychiatry outpatients. The pilot study uses a pre-post test design with two groups of 100 patients each from two clinics that serve primarily Latino patients. The group at the CHA clinic will serve as the "treatment" group. This group will receive the training modules and will be interviewed about their experience in care. The group at the clinic at Massachusetts General Hospital will serve as the "control" group. This group will be interviewed without first receiving the training. Outcomes for the groups will be compared to look for an effect. If the RQP training appears to have a positive affect on patients at CHA, then MGH patients will be offered the RQP training. By testing the effectiveness of this educational module, we hope to establish its usefulness as a means for the Cambridge Health Alliance to become even more patient-centered and to assist in the integration and institutionalization of patient empowerment/activation.

ELIGIBILITY:
Inclusion Criteria:

* Must be a mental health outpatient at selected clinics

Exclusion Criteria:

* Unable to verbalize or take verbal direction
* Unable to sit still in one place to participate in education modules
* Potentially violent towards others

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2004-08; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Patient activation | at 4, 6 and 8 weeks
Patient empowerment at 4, 6 and 8 weeks | at 4, 6 and 8 weeks
Retention in care at one year | at one year

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Alegria, PhD, Principal Investigator — Cambridge Health Alliance
Locations (2):
- United States (2):
  - Windsor Street Health Center, Cambridge, Massachusetts
  - MGH Chelsea Healthcare Center, Chelsea, Massachusetts